CLINICAL TRIAL: NCT05457530
Title: Effect of Modified, Rapid-start, DOR/3TC/TDF or DOR + FTC/TAF or BIC/FTC/TAF on Body Weight and Composition, Metabolic Risk Parameters, and Measures of Bone Strength in Treatment-Naïve Black and Hispanic Women With HIV-1 Infection
Brief Title: Doravirine and Weight Gain in Antiretroviral Naive
Acronym: DAWN
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to No/Low enrollment
Sponsor: Prism Health North Texas (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60160
Record Dates: First submitted 2022-04-15; First posted 2022-07-14 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Body Weight Changes; Human Immunodeficiency Virus; ART; Obesity; Minority Health; BMD; Metabolic Syndrome; Fasting
Keywords: Treatment Naive; African American Women; Hispanic Women; Fasting Glucose; Fasting Insuline; Negative pregnancy test; 18 years or older
MeSH Terms: conditions — Body Weight Changes; Acquired Immunodeficiency Syndrome; Obesity; Metabolic Syndrome; Fasting | interventions — Receptors, Opioid, delta; doravirine; emtricitabine tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (Active Comparator): Participants to receive DOR/3TC/TDF tablet once daily for 48 weeks
  Interventions: Drug: DOR/3TC/TDF
- Doravirine + Emtricitibine/Tenofovir alafenamide Fumerate (Active Comparator): Participants to receive DOR + FTC/TAF tablets once daily for 48 weeks
  Interventions: Combination Product: DOR + FTC/TAF
- Bictegravir/Emtricitibine/Tenofovir alafenamide (Active Comparator): Participants to receive BIC/FTC/TAF tablet once daily for 48 weeks
  Interventions: Drug: BIC/FTC/TAF

INTERVENTIONS:
Drug: DOR/3TC/TDF — 100 mg of doravirine (DOR), 300 mg of lamivudine (3TC), and 300 mg of TDF
  Other Names: Delstrigo
  Arms: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate
Combination Product: DOR + FTC/TAF — 100 mg of doravirine + 200 mg emtricitabine (FTC) and 25 mg of tenofovir alefenamide fumerate (TAF)
  Other Names: Pifeltro + Descovy
  Arms: Doravirine + Emtricitibine/Tenofovir alafenamide Fumerate
Drug: BIC/FTC/TAF — Bictegravir sodium 50 mg, emtricitabine 200mg, tenofovir alefenamide fumerate 25mg
  Other Names: Biktarvy
  Arms: Bictegravir/Emtricitibine/Tenofovir alafenamide

SUMMARY:
The purpose of this study is determine whether different antiretroviral therapy (ART) changes the effects on body fat and predict the weight change in Black and Hispanic females.

DETAILED DESCRIPTION:
Study is three-arm, open-label, randomized, interventional trial, in which all patients who are successfully enrolled will be randomized 1:1:1 to initiate ART therapy with Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate vs. Doravirine + Emtricitabine/Tenofovir Alefenamide, Bictegravir/Emtricitabine/Tenofovir Alafenamide. All patients will be followed or a total o 48 weeks.

.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* No prior exposure to antiretroviral therapy for >7 days prior to study entry;
* Plasma HIV1 RNA concentration >/=5000 copies/mL;
* CD4 T cell count >/=200 cells/µL.
* For persons capable of becoming pregnant, negative serum or urine pregnancy test within 45 days prior to entry
* Ability and willingness of participant or legal guardian/representative to provide informed consent

Exclusion Criteria:

* Evidence of resistance to DOR, TDF, 3TC/FTC or BIC.
* Creatinine clearance <60 mL/min
* Use of weight loss agents or plans to initiate weight loss program (diet or exercise-based)
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of BMI after Initiation of ART Therapy at Week 48 | Week 48
  Comparison of weight and height is collected prior to, and during ART to determine baseline and changes of BMI (kg/m2) on ART.
Change of BMI Category after Initiation of ART Therapy at Week 48 | Week 48
  Comparison of participants w/ >10% weight change in the study arms. BMI categories: underweight (<18.5) or normal weight (18.5 - 25) or overweight (25 - 30) or obese (>30); or from overweight to obese.
Change in Regional Lean and Body Mass | Week 48
  Whole body Dual-energy X-ray absorptiometry (DEXA) scan (Hologic, QDR 4500A) will measure changes between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Bedimo, Principal Investigator — Prism Health North Texas
Locations (1):
- Prism Health North Texas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No